CLINICAL TRIAL: NCT04220411
Title: A Phase I/IIa Open-Label, Dose-Escalation Study to Determine the Safety, Tolerability, and Efficacy of AR100DP1 in Healthy Subjects, and Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: A Study for AR100DP1 in Mild to Moderate Atopic Dermatitis (AD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the two AEs in Phase IIa study, recruiting was stopped for safety sake. The study was currently terminated.
Sponsor: Arjil Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AR100DP1-01
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Phase I: conventional 3+3 design of dose escalation Phase IIa: single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AR100DP1 (1.25%)_Phase I (Experimental): Subjects topically apply AR100DP1 twice per day with at least 4 hour interval. The daily dosage of 1.25% AR100DP1 topical administration is 31.25 mg/day (1.25% × 1,250 × 2 = 31.25).
  Interventions: Drug: AR100DP1
- AR100DP1 (2.5%)_Phase I (Experimental): Subjects topically apply AR100DP1 twice per day with at least 4 hour interval. The daily dosage of 2.5% AR100DP1 topical administration is 62.5 mg/day (2.5% × 1,250 × 2 = 62.5).
  Interventions: Drug: AR100DP1
- AR100DP1 (5%)_Phase I (Experimental): Subjects topically apply AR100DP1 twice per day with at least 4 hour interval. The daily dosage of 5% AR100DP1 topical administration is 125 mg/day (5% × 1,250 × 2 = 125).
  Interventions: Drug: AR100DP1
- AR100DP1 (5%)_Phase IIa (Experimental): Subjects topically apply AR100DP1 twice per day with at least 4 hour interval. The daily dosage of 5% AR100DP1 topical administration is 125 mg/day (5% × 1,250 × 2 = 125).
  Interventions: Drug: AR100DP1

INTERVENTIONS:
Drug: AR100DP1 — topical ointment

SUMMARY:
This is a Phase I/IIa Open-Label, Dose-Escalation Study to Determine the Safety, Tolerability, and Efficacy of AR100DP1 in Health Subjects, and Subjects with Mild to Moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
This phase I/IIa study will be composed of a Phase I study, which includes 14 days of treatment with AR100DP1 followed by 2 weeks of follow-up period to find the maximum tolerated dose (MTD) of AR100DP1 and a following single-arm Phase IIa study with 28 days of treatment followed by 2 weeks of follow-up period to evaluate the efficacy of AR100DP1 with the recommended Phase II dose (RP2D) in treating atopic dermatitis on target lesion. Target lesion area(s) is defined as one or multiple patches of lesion areas selected by the investigator for topical administration of AR100DP1. The size of target lesion area(s) is 0.5-5% body surface area (BSA) and the maximum is 750 cm2 (maximal treated area, inclusive) in this study. Eligible healthy subjects in Phase I will have the test skin area(s) of 750 cm2 from chest and abdomen. Eligible subjects with mild to moderate AD in Phase IIa will have target lesion area(s) selected by the investigator. The skin area treated with AR100DP1 will be recorded for AR100DP1 topical administration before dosing. AR100DP1 should be topically administered twice daily on the test skin area(s) of 750 cm2 of eligible healthy subjects for 14 days in Phase I study. The administration of AR100DP1 should be topically applied twice daily on target lesion area(s) (0.5-5% BSA, maximum as 750 cm2, inclusive) of eligible subjects with mild to moderate AD for 28 days in Phase IIa study.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

1. Dated and signed informed consent
2. Either gender, ≥ 20 years old (the legal age of consent majority is 20 years old in Taiwan)
3. Healthy subjects, who have no clinically relevant abnormalities, identified by medical history, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory tests
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures
5. Healthy skin on which reddening can be easily recognized in the area of the test fields, evaluated by the investigator
6. Subject of childbearing potential must agree to use abstinence to intercourse, or highly effective contraceptives from signing informed consent to 14 days after the last dose of study drug administration

At least two forms of effective birth control must be adopted for contraception, and one of which must be a barrier method. Acceptable forms include:

* Established use of oral, injected or implanted hormonal methods of contraception
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Barrier methods of contraception: condom (highly recommended with spermicide), or occlusive cap (diaphragm or cervical/vault caps)

Phase IIa:

1. Dated and signed informed consent
2. Either gender, ≥ 20 years old (the legal age of consent majority is 20 years old in Taiwan)
3. Confirmed clinical diagnosis of atopic dermatitis (based on the criteria of Hanifin and Rajka for AD)
4. With at least 0.5% body surface area (BSA) as target lesion area(s)
5. Clinical diagnosis of AD that has been clinically stable, which means the IGA score stays as 2 or 3 when evaluated for ≥ 4 weeks at the investigator's discretion prior to Screening Visit
6. With Investigator's Global Assessment (IGA) score of 2 (mild) or 3 (moderate) at screening
7. Subject of childbearing potential must agree to use abstinence to intercourse, or highly effective contraceptives from signing informed consent to 14 days after the last dose of study drug administration

At least two forms of effective birth control must be adopted for contraception, and one of which must be a barrier method. Acceptable forms include:

* Established use of oral, injected or implanted hormonal methods of contraception
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Barrier methods of contraception: condom (highly recommended with spermicide), or occlusive cap (diaphragm or cervical/vault caps)

Exclusion Criteria:

Phase I:

1. Subjects who have any visible skin disease at the application site which, in the opinion of the investigator, will interfere with the evaluation of the test site reaction
2. Subjects who have a history of AD, psoriasis and/or active AD/eczema
3. Subjects who have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site
4. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing)

Phase IIa:

1. Unstable or actively infected AD judged by the investigator.
2. Active or potentially recurrent dermatologic condition other than atopic dermatitis that may confound evaluation (e.g. fungal infection), judged by the investigator.
3. Received systemic medication including corticosteroid, immunosuppressant, anti-histamine, phototherapy, or other therapy, which could affect AD within 4 weeks before Screening. However, subjects are allowed to enter the study if subjects have been taking at least 2 weeks of fixed dose anti-histamine prior to Screening and this application does not affect the study judged by the investigator
4. Received topical medication including corticosteroid, immunosuppressant, anti-histamine, phototherapy, calcineurin inhibitors, or other therapy for AD on the target lesion area(s) within 1 week before Screening

   The following exclusion criteria are applied for all subjects in Phase I/IIa study:
5. Plan to receive immunosuppressive agents (including azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, cyclosporine), or systemic steroid with equivalent dosage higher than prednisolone 30 mg/day for more than 14 days at Screening
6. Unwilling or unable to comply with the criteria in Life Style Guidelines during the study
7. History of use of biologic therapy (including intravenous immunoglobulin) within 12 weeks or 5 half-lives (whichever is longer) prior to Screening
8. Received any other investigational drug within 4 weeks prior to Screening
9. Required or received systemic CYP3A4 inhibitors with strong potency within 1 week prior to screening, including but not limited to clarithromycin, itraconazole, nefazodone and atazanavir, evaluated by the investigator
10. Treatment for any type of cancer (except squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin, curatively treated with cryosurgery or surgical excision only) within 5 years before screening
11. Had surgery within 4 weeks prior to Screening Visit, or plan to have surgery during the study
12. Allergies requiring acute or chronic treatment at the investigator's discretion
13. Known hypersensitivity to any of the components of the study drug
14. Active clinically serious infection or history of human immunodeficiency virus (HIV) infection
15. Any of the following serum test abnormalities:

    * Total bilirubin > 1.5 × ULN
    * AST or ALT > 3.0 × ULN
    * Serum albumin < 2.5 g/dL
    * Creatinine > 1.5 × ULN
    * Any other ≥ Grade 2 (grading of vaccine clinical trials for Phase I and NCI-CTCAE v5.0 for Phase IIa) laboratory abnormality at baseline (other than those listed above)
16. With ongoing acute diseases or within the past 2 years serious medical conditions (e.g. concomitant illness) such as cardiovascular (e.g. New York Heart Association (NYHA) grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition (e.g. alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject
17. Female subject who is lactating or has positive urine pregnancy test at screening
18. Other conditions not suitable for participating in this study judged by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arjil Pharmaceuticals LLC., Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 subjects were screened in this study.
Pre-assignment Details: No screen failure occurred with final 17 eligible subjects.
Period: Overall Study
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Started | 6 | 3 | 6 | 2
Completed | 6 | 3 | 6 | 1
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Final Visit was Visit 6 (Day 29) for Phase I subjects, but Visit 8 (Day 43) for Phase II subjects. One subject in Phase II was early terminated at Visit 5.
Groups:
- AR100DP1 (5%)_Phase II: Subjects topically apply AR100DP1 twice per day with at least 4 hour interval. The daily dosage of 5% AR100DP1 topical administration is 125 mg/day (5% × 1,250 × 2 = 125).
- Total: Total of all reporting groups
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase II | Total
Number analyzed (Participants) | 6 | 3 | 6 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (4.07) | 26.7 (3.79) | 26.8 (0.98) | 29.0 (11.31) | 29.9 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 1 | 10
  Male | 3 | 1 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 6 | 2 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 6 | 3 | 6 | 2 | 17
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.3 (11.59) | 164.3 (8.50) | 164.3 (9.80) | 161.8 (5.94) | 165.4 (9.42)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 67.3 (10.19) | 60.1 (7.00) | 61.1 (16.70) | 78.7 (18.81) | 63.15 (13.55)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.63) | 22.5 (4.71) | 22.3 (4.35) | 29.9 (4.99) | 23.7 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With DLTs
Description: Phase I study included 14 days of treatment with AR100DP1, followed by 2 weeks of follow-up period to find the maximum tolerated dose (MTD) of AR100DP1.
  DLTs were defined as any adverse event (AE) ≥ Grade 2 (Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, issued by United States Food and Drug Administration in September 2007), that was considered to be causally related (possibly, probably, or definitely related) to AR100DP1 as judged by the investigator up to Day 29. The definition of Grade 5 (death related to AE) was added to this grading system as it was not defined in the guidance. (reported in the subsequent Primary Outcome Measure). MTD is defined as the highest dose level at which < 2 of 6 subjects experienced a dose-limiting toxicity (DLT).
Time Frame: up to Day 29 for each cohort in phase I
Population: All subjects received AR100DP1 at least 12 days with at least 85% of compliance.
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I
Number analyzed (Participants) | 6 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of AR100DP1
Description: Per protocol, MTD is defined as the highest dose level at which < 2 of 6 subjects experienced a dose-limiting toxicity (DLT).
  MTD was determined by testing increasing doses up to 125 mg/day via topical administration on AR100DP1_1.25%, 2.5%, and 5% groups with 3 to 6 subjects each.
  DLTs were defined as any adverse event (AE) ≥ Grade 2 (Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, issued by United States Food and Drug Administration in September 2007), that was considered to be causally related (possibly, probably, or definitely related) to AR100DP1 as judged by the investigator up to Day 29. The definition of Grade 5 (death related to AE) was added to this grading system as it was not defined in the guidance. (reported in the previous Primary Outcome Measure).
Time Frame: up to Day 29 for each cohort in phase I
Measure: Number; unit: mg/day
Groups:
- All Subjects in Phase I: All participants topically applied 1.25%, 2.5%, or 5% AR100DP1 twice daily at least 4-hour intervals.
  The daily dosages of 1.25%, 2.5%, and 5% AR100DP1 topical administration are 31.25 mg/day (1.25% × 1,250 × 2 = 31.25), 62.5 mg/day(2.5% × 1,250 × 2 = 62.5), and 125 mg/day (5% × 1,250 × 2 = 125), respectively.
Arm/Group | All Subjects in Phase I
Number analyzed (Participants) | 15
mg/day | 125

3. Primary Outcome: Percentage of Subjects With the Investigator's Global Assessment (IGA) Score of 0 or 1 on Day 29 (Phase IIa)
Description: The IGA is a 5-point scale that provides a global clinical assessment of AD severity based on an ordinal scale, scored by the investigator. The scores of IGA are 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (Severe).
Time Frame: Day 29 (Phase IIa)
Population: Efficacy analyses were conducted in phase IIa. Phase IIa was terminated early because of the safety issue. One subject in phase IIa was withdrawn from the study after Visit 6 (Day 29).
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
Participants
  Visit 1 (screening, Da -14~1) (Phase IIa) : Score 0 (clear) | 0
  Visit 1 (screening, Da -14~1) (Phase IIa) : Score 1 (almost clear) | 0
  Baseline (Phase IIa) : Score 0 (clear) | 0
  Baseline (Phase IIa) : Score 1 (almost clear) | 0
  Visit 6 (Day 29) (Phase IIa) : Score 0 (clear): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) : Score 0 (clear) | 0
  Visit 6 (Day 29) (Phase IIa) : Score 1 (almost clear): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) : Score 1 (almost clear) | 0

4. Secondary Outcome: Percentage of Subjects With the Investigator's Global Assessment (IGA) Score of 0 ~ 4 (Phase IIa)
Description: as for outcome 3
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
Participants
  Visit 1 (screening, Da -14~1) (Phase IIa): Score 0 (clear) | 0
  Visit 1 (screening, Da -14~1) (Phase IIa): Score 1 (almost clear) | 0
  Visit 1 (screening, Da -14~1) (Phase IIa): Score 2 (mild) | 1
  Visit 1 (screening, Da -14~1) (Phase IIa): Score 3 (moderate) | 1
  Visit 1 (screening, Da -14~1) (Phase IIa): Score 4 (severe) | 0
  Baseline (Phase IIa): Score 0 (clear) | 0
  Baseline (Phase IIa): Score 1 (almost clear) | 0
  Baseline (Phase IIa): Score 2 (mild) | 1
  Baseline (Phase IIa): Score 3 (moderate) | 1
  Baseline (Phase IIa): Score 4 (severe) | 0
  Visit 3 (Day 8) (Phase IIa): Score 0 (clear) | 0
  Visit 3 (Day 8) (Phase IIa): Score 1 (almost clear) | 0
  Visit 3 (Day 8) (Phase IIa): Score 2 (mild) | 2
  Visit 3 (Day 8) (Phase IIa): Score 3 (moderate) | 0
  Visit 3 (Day 8) (Phase IIa): Score 4 (severe) | 0
  Visit 4 (Day 15) (Phase IIa): Score 0 (clear) | 0
  Visit 4 (Day 15) (Phase IIa): Score 1 (almost clear) | 0
  Visit 4 (Day 15) (Phase IIa): Score 2 (mild) | 1
  Visit 4 (Day 15) (Phase IIa): Score 3 (moderate) | 0
  Visit 4 (Day 15) (Phase IIa): Score 4 (severe) | 1
  Visit 5 (Day 22) (Phase IIa): Score 0 (clear) | 0
  Visit 5 (Day 22) (Phase IIa): Score 1 (almost clear) | 0
  Visit 5 (Day 22) (Phase IIa): Score 2 (mild) | 1
  Visit 5 (Day 22) (Phase IIa): Score 3 (moderate) | 0
  Visit 5 (Day 22) (Phase IIa): Score 4 (severe) | 1
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa): Score 0 (clear) | 0
  Visit 6 (Day 29) (Phase IIa): Score 1 (almost clear) | 0
  Visit 6 (Day 29) (Phase IIa): Score 2 (mild) | 0
  Visit 6 (Day 29) (Phase IIa): Score 3 (moderate) | 0
  Visit 6 (Day 29) (Phase IIa): Score 4 (severe) | 1
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa): Score 0 (clear) | 0
  Visit 7 (Day 36) (Phase IIa): Score 1 (almost clear) | 0
  Visit 7 (Day 36) (Phase IIa): Score 2 (mild) | 1
  Visit 7 (Day 36) (Phase IIa): Score 3 (moderate) | 0
  Visit 7 (Day 36) (Phase IIa): Score 4 (severe) | 0
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa): Score 0 (clear) | 0
  Visit 8 (Day 43) (Phase IIa): Score 1 (almost clear) | 1
  Visit 8 (Day 43) (Phase IIa): Score 2 (mild) | 0
  Visit 8 (Day 43) (Phase IIa): Score 3 (moderate) | 0
  Visit 8 (Day 43) (Phase IIa): Score 4 (severe) | 0

5. Secondary Outcome: Change From Baseline in Pruritus Numerical Rating Scale (NRS) of Itch Level on Target Lesions
Description: The pruritus NRS is comprised itch level grading from the numbers 0 ("no itch") to 10 ("worst imaginable itch"). Subjects are asked to rate the intensity of their itch by visits.
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
score on a scale
  Visit 2 (Day 1) (Phase IIa) | 6.50 (0.707)
  Visit 3 (Day 8) (Phase IIa) | 2.00 (0.000)
  Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -4.50 (0.707)
  Visit 4 (Day 15) (Phase IIa) | 5.50 (6.364)
  Visit 4 (Day 15)-Visit 2 (Day 1) | -1.00 (5.657)
  Visit 5 (Day 22) (Phase IIa) | 7.50 (3.536)
  Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | 1.00 (2.828)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) | 6.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | -5.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | -6.00 (NA) — It was not applicable due to only 1 subject's data.

6. Secondary Outcome: Change of IgE Compared to Baseline (Day 1)
Time Frame: Day 15 and 29 (Phase IIa)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
IU/mL
  Visit 2 (Day 1) (Phase IIa) | 7.15 (0.198)
  Visit 4 (Day 15) (Phase IIa) | 7.17 (0.091)
  Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | 0.02 (0.106)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) | 7.09 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 0.08 (NA) — It was not applicable due to only 1 subject's data.

7. Secondary Outcome: Fold Change of IL-4 Compared to Baseline (Day 1 )
Time Frame: Day 15 and 29 (Phase IIa)
Population: No source data was collected for IL-4 in this study.
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Signs of Atopic Dermatitis (Erythema, Edema, Excoriation and Lichenification) on Target Lesions
Description: 4 symptoms of atopic dermatitis (erythema, edema, excoriation and lichenification) will be evaluated on all target lesions and graded from 0 to 3 (none, mild, moderate and severe, respectively), with half points allowed
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
score on a scale
  Erythema: Visit 2 (Day 1) (Phase IIa) | 1.50 (0.707)
  Erythema: Visit 3 (Day 8) (Phase IIa) | 0.75 (1.061)
  Erythema: Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -0.75 (0.354)
  Erythema: Visit 4 (Day 15) (Phase IIa) | 1.50 (2.121)
  Erythema: Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | 0.00 (1.414)
  Erythema: Visit 5 (Day 22) (Phase IIa) | 2.00 (1.414)
  Erythema: Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | 0.50 (0.707)
  Erythema: Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 6 (Day 29) (Phase IIa) | 2.5 (NA) — It was not applicable due to only 1 subject's data.
  Erythema: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 1.5 (NA) — It was not applicable due to only 1 subject's data.
  Erythema: Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 7 (Day 36) (Phase IIa) | 2.00 (NA) — It was not applicable due to only 1 subject's data.
  Erythema: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Erythema: Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 8 (Day 43) (Phase IIa) | 0.50 (NA) — It was not applicable due to only 1 subject's data.
  Erythema: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Erythema: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | -0.50 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 2 (Day 1) (Phase IIa) | 1.00 (0.000)
  Edema: Visit 3 (Day 8) (Phase IIa) | 0.75 (0.354)
  Edema: Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -0.25 (0.354)
  Edema: Visit 4 (Day 15) (Phase IIa) | 1.25 (1.768)
  Edema: Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | 0.25 (1.768)
  Edema: Visit 5 (Day 22) (Phase IIa) | 2.00 (1.414)
  Edema: Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | 1.00 (1.414)
  Edema: Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 6 (Day 29) (Phase IIa) | 2.00 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 7 (Day 36) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 8 (Day 43) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Edema: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Edema: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | -1.00 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 2 (Day 1) (Phase IIa) | 1.25 (1.061)
  Excoriation: Visit 3 (Day 8) (Phase IIa) | 0.75 (0.354)
  Excoriation: Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -0.50 (0.707)
  Excoriation: Visit 4 (Day 15) (Phase IIa) | 0.25 (0.354)
  Excoriation: Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | -1.00 (0.707)
  Excoriation: Visit 5 (Day 22) (Phase IIa) | 0.50 (0.000)
  Excoriation: Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | -0.75 (1.061)
  Excoriation: Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 6 (Day 29) (Phase IIa) | 3.00 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 2.50 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 7 (Day 36) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | 0.50 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 8 (Day 43) (Phase IIa) | 0.50 (NA) — It was not applicable due to only 1 subject's data.
  Excoriation: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Excoriation: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 2 (Day 1) (Phase IIa) | 1.75 (0.354)
  Lichenification: Visit 3 (Day 8) (Phase IIa) | 1.00 (0.000)
  Lichenification: Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -0.75 (0.354)
  Lichenification: Visit 4 (Day 15) (Phase IIa) | 0.75 (0.354)
  Lichenification: Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | -1.00 (0.707)
  Lichenification: Visit 5 (Day 22) (Phase IIa) | 0.75 (0.354)
  Lichenification: Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | -1.00 (0.707)
  Lichenification: Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 6 (Day 29) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | -1.00 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 7 (Day 36) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | -1.00 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 8 (Day 43) (Phase IIa) | 0.50 (NA) — It was not applicable due to only 1 subject's data.
  Lichenification: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Lichenification: Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | -1.50 (NA) — It was not applicable due to only 1 subject's data.

9. Secondary Outcome: Change From Baseline in the Total Score of Patient-Oriented Eczema Measure (POEM)
Description: POEM is a validated, patient-derived assessment measure for monitoring atopic eczema severity , available at the HOME (Harmonising Outcome Measures for Eczema) group. It contains seven symptoms of AD on 5-point (0 to 4) scale with total score 0 to 28 during the study.
  A higher score means a worse outcome, whereas a lower score is a better outcome.
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
score on a scale
  Visit 2 (Day 1) (Phase IIa) | 13.50 (4.950)
  Visit 3 (Day 8) (Phase IIa) | 4.50 (0.707)
  Visit 3 (Day 8)-Visit 2 (Day 1) (Phase IIa) | -9.00 (4.243)
  Visit 4 (Day 15) (Phase IIa) | 4.50 (4.950)
  Visit 4 (Day 15)-Visit 2 (Day 1) (Phase IIa) | -9.00 (0.000)
  Visit 5 (Day 22) (Phase IIa) | 7.00 (2.828)
  Visit 5 (Day 22)-Visit 2 (Day 1) (Phase IIa) | -6.50 (7.778)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) | 25.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29)-Visit 2 (Day 1) (Phase IIa) | 15.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa) | 11.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36)-Visit 2 (Day 1) (Phase IIa) | 1.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa) | 0.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43)-Visit 2 (Day 1) (Phase IIa) | -10.00 (NA) — It was not applicable due to only 1 subject's data.

10. Secondary Outcome: Number of Subjects With AE and SAE
Time Frame: Day -14 to 29 (Phase I); Day -14 to 43 (Phase IIa)
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
Participants
  AE | 1 | 0 | 2 | 2
  Treatment-related AE | 0 | 0 | 1 | 2
  DLT | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 1
  SUSAR | 0 | 0 | 0 | 1
  Death | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Vital Signs (Systolic Blood Pressure)
Description: Vital signs measurement will consist of systolic/diastolic blood pressure, respiratory rate, pulse rate or heart rate, and body temperature.
Time Frame: Day 1 to 29 (Phase I); Day 1 to 43 (Phase IIa)
Population: Final visit was Visit 6 (Day 29) for Phase I subjects, but Visit 8 (Day 43) for Phase II subjects. Phase IIa was terminated early because of the safety issue. One subject in phase IIa was withdrawn from the study after Visit 6 (Day 29).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
mmHg
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I) | 104.17 (5.037) | 115.67 (12.662) | 118.67 (7.090) |
  Baseline (Day -14~ Day 1; Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Day -14~ Day 1; Phase I) | 116.33 (11.605) | 112.67 (11.150) | 115.50 (13.157) |
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 114.50 (9.503) | 116.00 (7.211) | 109.33 (13.471) |
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I) | -1.83 (8.727) | 3.33 (5.686) | -6.17 (16.810) |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 111.83 (11.143) | 121.33 (16.803) | 111.00 (7.563) |
  Visit 3 (Day 8) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) - Baseline (Phase I) | -4.50 (6.686) | 8.67 (27.006) | -4.50 (11.640) |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 116.00 (7.589) | 112.00 (14.731) | 112.83 (13.167) |
  Visit 4 (Day 15) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) - Baseline (Phase I) | -0.33 (9.309) | -0.67 (18.502) | -2.67 (11.448) |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 109.50 (10.654) | 122.67 (5.686) | 112.83 (9.109) |
  Visit 5 (Day 22) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) - Baseline (Phase I) | -6.83 (3.189) | 10.00 (9.165) | -2.67 (13.530) |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 118.17 (9.988) | 122.33 (2.887) | 108.67 (8.869) |
  Visit 6 (Day 29) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) - Baseline (Phase I) | 1.83 (9.065) | 9.67 (12.423) | -6.83 (11.652) |
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa) |  |  |  | 130.50 (24.749)
  Baseline (Day -14~ Day 1; Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Day -14~ Day 1; Phase IIa) |  |  |  | 130.00 (29.698)
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 136.00 (33.941)
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa) |  |  |  | 6.00 (4.243)
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 145.00 (32.527)
  Visit 3 (Day 8) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) - Baseline (Phase IIa) |  |  |  | 15.00 (2.828)
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 127.00 (11.314)
  Visit 4 (Day 15) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) - Baseline (Phase IIa) |  |  |  | -3.00 (18.385)
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 127.00 (19.799)
  Visit 5 (Day 22) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) - Baseline (Phase IIa) |  |  |  | -3.00 (9.899)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 149.00 (NA) — It was not applicable due to only 1 subject's data
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) |  |  |  | -2.00 (NA) — It was not applicable due to only 1 subject's data
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 142.00 (NA) — It was not applicable due to only 1 subject's data
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) |  |  |  | -9.00 (NA) — It was not applicable due to only 1 subject's data
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 129.00 (NA) — It was not applicable due to only 1 subject's data
  Visit 8 (Day 43) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) - Baseline (Phase IIa) |  |  |  | -22.00 (NA) — It was not applicable due to only 1 subject's data

12. Secondary Outcome: Number of Subjects With Physical Examination Abnormalities
Description: Physical examination will include the following items: general appearance, skin, eyes, ears, nose, throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological and others.
Time Frame: Day -14 to 29 (Phase I); Day -14 to 43 (Phase IIa)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
Participants
  Visit 1 (Screening) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening) (Phase I) | 0 | 0 | 0 | 0
  Visit 2 (Day 1) : before IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : before IP Administration (Phase I) | 0 | 0 | 0 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 0 | 0 | 0 | 0
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 0 | 0 | 0 | 0
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 1 | 0 | 0 | 0
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 1 | 0 | 1 |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 1 | 0 | 1 |
  Visit 1 (Screening) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening) (Phase IIa) |  |  |  | 0
  Visit 2 (Day 1) : before IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : before IP Administration (Phase IIa) |  |  |  | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 0
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 1
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 1
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 1
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 1
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 1

13. Secondary Outcome: Number of Subjects With 12-lead ECG Abnormalities
Description: ECG will be evaluated by the investigators and noted as "Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical significant (CS)"
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29 (Phase I); Day 1, Day 8, Day 15, Day 22, Day 29, Day 43 (Phase IIa)
Population: Final visit was Visit 6 (Day 29) for Phase I subjects, but Visit 8 (Day 43) for Phase II subjects.Phase IIa was terminated early because of the safety issue. One subject in phase IIa was withdrawn from the study after Visit 6 (Day 29).
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
Participants
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): Normal | 1 | 1 | 4 |
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): NCS | 5 | 2 | 2 |
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): CS (Medical History) | 0 | 0 | 0 |
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): CS (Adverse Event) | 0 | 0 | 0 |
  Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Phase I): Normal | 2 | 1 | 3 | 0
  Baseline (Phase I): NCS | 4 | 2 | 3 | 0
  Baseline (Phase I): CS (Medical History) | 0 | 0 | 0 | 0
  Baseline (Phase I): CS (Adverse Event) | 0 | 0 | 0 | 0
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I): Normal | 3 | 2 | 3 |
  Visit 3 (Day 8) (Phase I): NCS | 3 | 1 | 3 |
  Visit 3 (Day 8) (Phase I): CS (Medical History) | 0 | 0 | 0 | 0
  Visit 3 (Day 8) (Phase I): CS (Adverse Event) | 0 | 0 | 0 | 0
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I): Normal | 4 | 0 | 2 | 0
  Visit 4 (Day 15) (Phase I): NCS | 2 | 3 | 4 | 0
  Visit 4 (Day 15) (Phase I): CS (Medical History) | 0 | 0 | 0 | 0
  Visit 4 (Day 15) (Phase I): CS (Adverse Event) | 0 | 0 | 0 | 0
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I): Normal | 3 | 1 | 2 |
  Visit 5 (Day 22) (Phase I): NCS | 3 | 2 | 4 | 0
  Visit 5 (Day 22) (Phase I): CS (Medical History) | 0 | 0 | 0 | 0
  Visit 5 (Day 22) (Phase I): CS (Adverse Event) | 0 | 0 | 0 | 0
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I): Normal | 1 | 0 | 2 |
  Visit 6 (Day 29) (Phase I): NCS | 5 | 3 | 4 | 0
  Visit 6 (Day 29) (Phase I): CS (Medical History) | 0 | 0 | 0 | 0
  Visit 6 (Day 29) (Phase I): CS (Adverse Event) | 0 | 0 | 0 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): Normal |  |  |  | 1
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): NCS |  |  |  | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): CS (Medical History) |  |  |  | 1
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Phase IIa): Normal |  |  |  | 1
  Baseline (Phase IIa): NCS |  |  |  | 1
  Baseline (Phase IIa): CS (Medical History) |  |  |  | 0
  Baseline (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa): Normal |  |  |  | 1
  Visit 3 (Day 8) (Phase IIa): NCS |  |  |  | 1
  Visit 3 (Day 8) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 3 (Day 8) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa): Normal |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): NCS |  |  |  | 2
  Visit 4 (Day 15) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa): Normal |  |  |  | 2
  Visit 5 (Day 22) (Phase IIa): NCS |  |  |  | 0
  Visit 5 (Day 22) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 5 (Day 22) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa): Normal |  |  |  | 1
  Visit 6 (Day 29) (Phase IIa): NCS |  |  |  | 0
  Visit 6 (Day 29) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 6 (Day 29) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa): Normal |  |  |  | 1
  Visit 7 (Day 36) (Phase IIa): NCS |  |  |  | 0
  Visit 7 (Day 36) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 7 (Day 36) (Phase IIa): CS (Adverse Event) |  |  |  | 0
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa): Normal |  |  |  | 1
  Visit 8 (Day 43) (Phase IIa): NCS |  |  |  | 0
  Visit 8 (Day 43) (Phase IIa): CS (Medical History) |  |  |  | 0
  Visit 8 (Day 43) (Phase IIa): CS (Adverse Event) |  |  |  | 0

14. Secondary Outcome: Number of Subjects With Clinically Significant Laboratory Abnormalities (Hematology)
Description: Laboratory tests include hematology (hemoglobin, hematocrit, RBC, platelet, WBC with different counts), biochemistry (total bilirubin, AST, ALT, serum creatinine and albumin)
Time Frame: Day 8 to Day 29 (Phase I); Day 8 to Day 43 (Phase IIa)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
Participants
  Visit 1 (Screening) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening) (Phase I) | 0 | 0 | 0 | 0
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 0 | 0 | 0 | 0
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 0 | 0 | 0 | 0
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 0 | 0 | 0 | 0
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 0 | 0 | 0 | 0
  Visit 1 (Screening) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening) (Phase IIa) |  |  |  | 0
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 0
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 1
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 0
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 0
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 0

15. Secondary Outcome: Change From Baseline in Vital Signs (Diastolic Blood Pressure)
Description: as for outcome 11
Time Frame: Day 1 to 29 (Phase I); Day 1 to 43 (Phase IIa)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
mmHg
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I) | 69.00 (7.537) | 76.33 (9.713) | 71.83 (7.139) |
  Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Phase I) | 66.17 (7.167) | 69.00 (9.539) | 72.00 (11.900) |
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 68.00 (3.950) | 69.33 (7.572) | 71.00 (9.209) |
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I) | 1.83 (8.329) | 0.33 (3.215) | -1.00 (12.759) |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 72.83 (6.555) | 77.00 (6.245) | 72.17 (5.672) |
  Visit 3 (Day 8) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) - Baseline (Phase I) | 6.67 (7.257) | 8.00 (9.539) | 0.17 (12.449) |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 74.83 (5.456) | 75.33 (10.408) | 70.17 (3.430) |
  Visit 4 (Day 15) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) - Baseline (Phase I) | 8.67 (7.737) | 6.33 (6.658) | -1.83 (9.042) |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 73.00 (6.986) | 63.67 (2.517) | 68.33 (6.314) |
  Visit 5 (Day 22) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) - Baseline (Phase I) | 6.83 (11.566) | -5.33 (7.095) | -3.67 (6.250) |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 72.83 (8.864) | 76.33 (10.263) | 70.00 (6.870) |
  Visit 6 (Day 29) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) - Baseline (Phase I) | 6.67 (13.779) | 7.33 (19.757) | -2.00 (7.925) |
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa) |  |  |  | 77.50 (19.092)
  Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Phase IIa) |  |  |  | 88.50 (27.577)
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 88.00 (31.113)
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa) |  |  |  | -0.50 (3.536)
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 91.50 (31.820)
  Visit 3 (Day 8) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) - Baseline (Phase IIa) |  |  |  | 3.00 (4.243)
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 85.00 (12.728)
  Visit 4 (Day 15) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) - Baseline (Phase IIa) |  |  |  | -3.50 (14.849)
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 78.00 (12.728)
  Visit 5 (Day 22) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) - Baseline (Phase IIa) |  |  |  | -10.50 (14.849)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 90.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) |  |  |  | -18.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 86.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) |  |  |  | -22.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 82.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) - Baseline (Phase IIa) |  |  |  | -26.00 (NA) — It was not applicable due to only 1 subject's data.

16. Secondary Outcome: Change From Baseline in Vital Signs (Pulse Rate)
Description: as for outcome 11
Time Frame: Day 1 to 29 (Phase I); Day 1 to 43 (Phase IIa)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
beats/min
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I) | 68.33 (6.439) | 74.00 (6.083) | 72.67 (8.189) |
  Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Phase I) | 75.50 (11.041) | 73.67 (1.528) | 76.33 (11.587) |
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 68.33 (6.470) | 71.33 (3.215) | 72.17 (7.278) |
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I) | -7.17 (5.776) | -2.33 (3.512) | -4.17 (10.666) |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 71.33 (9.004) | 91.00 (5.000) | 74.00 (9.143) |
  Visit 3 (Day 8) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) - Baseline (Phase I) | -4.17 (5.193) | 17.33 (6.506) | -2.33 (7.033) |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 69.50 (10.035) | 77.33 (9.452) | 72.83 (9.704) |
  Visit 4 (Day 15) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) - Baseline (Phase I) | -6.00 (5.692) | 3.67 (9.609) | -3.50 (5.822) |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 68.17 (7.679) | 68.00 (10.392) | 75.50 (4.231) |
  Visit 5 (Day 22) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) - Baseline (Phase I) | -7.33 (12.848) | -5.67 (10.214) | -0.83 (14.743) |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 71.00 (8.438) | 73.33 (13.317) | 75.50 (7.740) |
  Visit 6 (Day 29) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) - Baseline (Phase I) | -4.50 (12.865) | -0.33 (13.577) | -0.83 (12.416) |
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa) |  |  |  | 77.00 (14.142)
  Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Phase IIa) |  |  |  | 81.50 (3.536)
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 79.50 (3.536)
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa) |  |  |  | -2.00 (0.000)
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 81.50 (4.950)
  Visit 3 (Day 8) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) - Baseline (Phase IIa) |  |  |  | 0.00 (8.485)
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 78.00 (8.485)
  Visit 4 (Day 15) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) - Baseline (Phase IIa) |  |  |  | -3.50 (12.021)
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 84.50 (0.707)
  Visit 5 (Day 22) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) - Baseline (Phase IIa) |  |  |  | 3.00 (4.243)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 89.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) |  |  |  | 10.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 85.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) |  |  |  | 6.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 94.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) - Baseline (Phase IIa) |  |  |  | 15.00 (NA) — It was not applicable due to only 1 subject's data.

17. Secondary Outcome: Change From Baseline in Vital Signs (Respiration Rate)
Description: as for outcome 11
Time Frame: Day 1 to 29 (Phase I); Day 1 to 43 (Phase IIa)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
breaths/min
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I) | 13.33 (2.066) | 13.33 (1.155) | 13.33 (1.033) |
  Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Phase I) | 14.00 (1.789) | 12.67 (1.155) | 13.50 (1.225) |
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 12.33 (0.816) | 12.67 (1.155) | 13.17 (0.983) |
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I) | -1.67 (1.966) | 0.00 (2.000) | -0.33 (1.862) |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 13.00 (1.095) | 13.33 (1.155) | 14.17 (1.169) |
  Visit 3 (Day 8) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) - Baseline (Phase I) | -1.00 (1.095) | 0.67 (1.155) | 0.67 (1.751) |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 13.67 (1.506) | 12.67 (1.155) | 12.83 (0.983) |
  Visit 4 (Day 15) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) - Baseline (Phase I) | -0.33 (2.658) | 0.00 (0.000) | -0.67 (1.966) |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 13.00 (1.095) | 13.33 (1.155) | 13.67 (1.033) |
  Visit 5 (Day 22) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) - Baseline (Phase I) | -1.00 (1.673) | 0.67 (1.155) | 0.17 (1.941) |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 13.83 (0.408) | 12.67 (1.155) | 13.17 (0.983) |
  Visit 6 (Day 29) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) - Baseline (Phase I) | -0.17 (2.041) | 0.00 (0.000) | -0.33 (1.366) |
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa) |  |  |  | 16.00 (1.414)
  Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Phase IIa) |  |  |  | 15.50 (2.121)
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 15.50 (2.121)
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa) |  |  |  | 0.00 (0.000)
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 15.50 (2.121)
  Visit 3 (Day 8) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) - Baseline (Phase IIa) |  |  |  | 0.00 (0.000)
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 15.50 (2.121)
  Visit 4 (Day 15) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) - Baseline (Phase IIa) |  |  |  | 0.00 (0.000)
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 14.50 (3.536)
  Visit 5 (Day 22) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) - Baseline (Phase IIa) |  |  |  | -1.00 (1.414)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 13.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) |  |  |  | -1.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 12.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) |  |  |  | -2.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 12.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) - Baseline (Phase IIa) |  |  |  | -2.00 (NA) — It was not applicable due to only 1 subject's data.

18. Secondary Outcome: Change From Baseline in Vital Signs (Body Temperature)
Description: as for outcome 11
Time Frame: Day 1 to 29 (Phase I); Day 1 to 43 (Phase IIa)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: degree C
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
degree C
  Visit 1 (Screening, Day -14 ~ -1) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening, Day -14 ~ -1) (Phase I) | 36.30 (0.155) | 36.20 (0.200) | 36.13 (0.234) |
  Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Baseline (Phase I) | 36.28 (0.232) | 36.20 (0.400) | 36.35 (0.315) |
  Visit 2 (Day 1) : 30M after IP Administration (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration (Phase I) | 36.30 (0.110) | 36.23 (0.321) | 36.10 (0.303) |
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase I) | 0.02 (0.248) | 0.03 (0.473) | -0.25 (0.532) |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 36.30 (0.276) | 36.33 (0.231) | 36.17 (0.339) |
  Visit 3 (Day 8) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) - Baseline (Phase I) | 0.02 (0.376) | 0.13 (0.231) | -0.18 (0.204) |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 36.35 (0.362) | 36.07 (0.289) | 36.10 (0.297) |
  Visit 4 (Day 15) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) - Baseline (Phase I) | 0.07 (0.441) | -0.13 (0.493) | -0.25 (0.302) |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 36.40 (0.385) | 36.63 (0.153) | 36.10 (0.374) |
  Visit 5 (Day 22) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) - Baseline (Phase I) | 0.12 (0.515) | 0.43 (0.252) | -0.25 (0.476) |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 36.52 (0.360) | 36.53 (0.379) | 35.9 (0.141) |
  Visit 6 (Day 29) - Baseline (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) - Baseline (Phase I) | 0.23 (0.455) | 0.33 (0.737) | -0.45 (0.409) |
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening, Day -14 ~ -1) (Phase IIa) |  |  |  | 36.65 (0.071)
  Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Baseline (Phase IIa) |  |  |  | 36.25 (0.495)
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration (Phase IIa) |  |  |  | 36.30 (0.424)
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 2 (Day 1) : 30M after IP Administration - Baseline (Phase IIa) |  |  |  | 0.05 (0.071)
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 36.25 (0.495)
  Visit 3 (Day 8) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) - Baseline (Phase IIa) |  |  |  | 0.00 (0.000)
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 36.45 (0.212)
  Visit 4 (Day 15) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) - Baseline (Phase IIa) |  |  |  | 0.20 (0.283)
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 36.55 (0.071)
  Visit 5 (Day 22) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) - Baseline (Phase IIa) |  |  |  | 0.30 (0.424)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 36.00 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) |  |  |  | 0.10 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 36.40 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) |  |  |  | 0.50 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 36.60 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) - Baseline (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) - Baseline (Phase IIa) |  |  |  | 0.70 (NA) — It was not applicable due to only 1 subject's data.

19. Secondary Outcome: Number of Subjects With Clinically Significant Laboratory Abnormalities (Biochemistry)
Description: as for outcome 14
Time Frame: Day 8 to Day 29 (Phase I); Day 8 to Day 43 (Phase IIa)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 6 | 3 | 6 | 2
Participants
  Visit 1 (Screening) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 1 (Screening) (Phase I) | 0 | 0 | 0 |
  Visit 3 (Day 8) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 3 (Day 8) (Phase I) | 0 | 0 | 0 |
  Visit 4 (Day 15) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 4 (Day 15) (Phase I) | 0 | 0 | 0 |
  Visit 5 (Day 22) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 5 (Day 22) (Phase I) | 0 | 0 | 0 |
  Visit 6 (Day 29) (Phase I): number analyzed (Participants) | 6 | 3 | 6 | 0
  Visit 6 (Day 29) (Phase I) | 0 | 0 | 0 |
  Visit 1 (Screening) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 1 (Screening) (Phase IIa) |  |  |  | 0
  Visit 3 (Day 8) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 3 (Day 8) (Phase IIa) |  |  |  | 0
  Visit 4 (Day 15) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 4 (Day 15) (Phase IIa) |  |  |  | 0
  Visit 5 (Day 22) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 2
  Visit 5 (Day 22) (Phase IIa) |  |  |  | 0
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 6 (Day 29) (Phase IIa) |  |  |  | 0
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 7 (Day 36) (Phase IIa) |  |  |  | 0
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 0 | 0 | 0 | 1
  Visit 8 (Day 43) (Phase IIa) |  |  |  | 0

20. Secondary Outcome: Percentage of Subjects Achieving the Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) on Day 8, Day 15, Day 22, Day 36 and Day 43 (Phase IIa)
Description: as for outcome 3
Time Frame: Day 8, Day 15, Day 22, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
Participants
  Visit 1 (screening, Da -14~1) (Phase IIa) : Score 0 (clear) | 0
  Visit 1 (screening, Da -14~1) (Phase IIa) : Score 1 (almost clear) | 0
  Baseline (Phase IIa) : Score 0 (clear) | 0
  Baseline (Phase IIa) : Score 1 (almost clear) | 0
  Visit 3 (Day 8) (Phase IIa) : Score 0 (clear) | 0
  Visit 3 (Day 8) (Phase IIa) : Score 1 (almost clear) | 0
  Visit 4 (Day 15) (Phase IIa) : Score 0 (clear) | 0
  Visit 4 (Day 15) (Phase IIa) : Score 1 (almost clear) | 0
  Visit 5 (Day 22) (Phase IIa) : Score 0 (clear) | 0
  Visit 5 (Day 22) (Phase IIa) : Score 1 (almost clear) | 0
  Visit 7 (Day 36) (Phase IIa) : Score 0 (clear): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa) : Score 0 (clear) | 0
  Visit 7 (Day 36) (Phase IIa) : Score 1 (almost clear): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa) : Score 1 (almost clear) | 0
  Visit 8 (Day 43) (Phase IIa) : Score 0 (clear): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa) : Score 0 (clear) | 0
  Visit 8 (Day 43) (Phase IIa) : Score 1 (almost clear): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa) : Score 1 (almost clear) | 0

21. Secondary Outcome: Change From Baseline of Target Lesion Area(s) on Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 (Phase IIa)
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 36 and Day 43 (Phase IIa)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AR100DP1 (5%)_Phase IIa
Number analyzed (Participants) | 2
cm^2
  Visit 1 (screening, Da -14~1) (Phase IIa) | 159.16 (7.870)
  Baseline (Phase IIa) | 157.93 (10.805)
  Visit 3 (Day 8) (Phase IIa) | 113.21 (19.757)
  Visit 3 (Day 8) - Baseline (Phase IIa) | -44.72 (8.952)
  Visit 4 (Day 15) (Phase IIa) | 287.84 (349.891)
  Visit 4 (Day 15) - Baseline (Phase IIa) | 129.91 (339.086)
  Visit 5 (Day 22) (Phase IIa) | 540.09 (145.593)
  Visit 5 (Day 22) - Baseline (Phase IIa) | 382.16 (134.789)
  Visit 6 (Day 29) (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) (Phase IIa) | 291.18 (NA) — It was not applicable due to only 1 subject's data.
  Visit 6 (Day 29) - Baseline (Phase IIa): number analyzed (Participants) | 1
  Visit 6 (Day 29) - Baseline (Phase IIa) | 140.89 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36) (Phase IIa) | 121.45 (NA) — It was not applicable due to only 1 subject's data.
  Visit 7 (Day 36) - Baseline (Phase IIa): number analyzed (Participants) | 1
  Visit 7 (Day 36) - Baseline (Phase IIa) | -28.84 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43) (Phase IIa) | 46.78 (NA) — It was not applicable due to only 1 subject's data.
  Visit 8 (Day 43) -Baseline (Phase IIa): number analyzed (Participants) | 1
  Visit 8 (Day 43) -Baseline (Phase IIa) | -103.51 (NA) — It was not applicable due to only 1 subject's data.

ADVERSE EVENTS:
Time Frame: Day -14 to 29 (Phase I); Day -14 to 43 (Phase IIa)
Arm/Group | AR100DP1 (1.25%)_Phase I | AR100DP1 (2.5%)_Phase I | AR100DP1 (5%)_Phase I | AR100DP1 (5%)_Phase II
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 1/2
Other Adverse Events (participants affected / at risk) | 1/6 | 0/3 | 2/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR100DP1 (1.25%)_Phase I (N=6) | AR100DP1 (2.5%)_Phase I (N=3) | AR100DP1 (5%)_Phase I (N=6) | AR100DP1 (5%)_Phase II (N=2)
Irritant contact dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR100DP1 (1.25%)_Phase I (N=6) | AR100DP1 (2.5%)_Phase I (N=3) | AR100DP1 (5%)_Phase I (N=6) | AR100DP1 (5%)_Phase II (N=2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site dermatitis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT04220411/Prot_SAP_000.pdf